CLINICAL TRIAL: NCT01489358
Title: VRC 311: A Phase 1 Open Label, Dose-Escalation Clinical Trial to Evaluate the Safety and Immunogenicity of a Virus-Like Particle (VLP) Chikungunya Vaccine, VRC-CHKVLP059-00-VP, in Healthy Adults
Brief Title: Chikungunya Virus Vaccine Trial in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 120041; 12-I-0041 (Other: NIH)
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-03

CONDITIONS: Viral Vaccines; Chikungunya Fever; Chikungunya Virus Infection
Keywords: Vaccine-Mediated Protection; Antibody Response; Chikungunya Virus; Immune Response; Healthy Volunteer; Humoral Inmunity; Virus-like Particles
MeSH Terms: conditions — Chikungunya Fever

ARMS (3):
- Group 1 (Experimental): Group 1 will receive three IM injections of VRC-CHKVLP059-00-VP (at weeks 0,4, and 20) at a dose of 10 mcg.
  Interventions: Biological: VRC-CHKVLP059-00-VP
- Group 2 (Experimental): Group 2 will receive three IM injections of VRC-CHKVLP059-00-VP (at weeks 0,4, and 20) at a dose of 20 mcg.
  Interventions: Biological: VRC-CHKVLP059-00-VP
- Group 3 (Experimental): Group 3 will receive three IM injections of VRC-CHKVLP059-00-VP (at weeks 0,4, and 20) at a dose of 40 mcg.
  Interventions: Biological: VRC-CHKVLP059-00-VP

INTERVENTIONS:
Biological: VRC-CHKVLP059-00-VP — VRC-CHKVLP059-00-VP is a VLP vaccine that consists of the E1, E2 and capsid proteins of the Chikungunya Virus

SUMMARY:
Background:

- Chikungunya virus (CHIKV) is transmitted by mosquitoes. It can cause fever, headache, muscle pain, fatigue, and joint pain. The disease usually does not cause death. But the joint pain, which may be directly related to the infecting virus, may be severe and last for several months. CHIKV outbreaks are most common in Africa, India, and Asia. A new experimental vaccine for CHIKV has been developed, and researchers are testing it in healthy adults. Participants cannot develop CHIKV from this vaccine.

Objectives:

- To test the safety and effectiveness of a Chikungunya virus vaccine.

Eligibility:

- Healthy individuals between 18 and 50 years of age.

Design:

* This study, including vaccine doses and followup tests, will last about 44 weeks. Participants will have three vaccination visits, six followup clinic visits, and three telephone contacts during this study. Vaccination visits will take about 4 hours. Most other clinic visits will usually take 2 hours. The telephone contacts will take about 15 minutes.
* Participants will be screened with a physical exam and medical history. Blood samples will also be collected.
* Participants will be assigned to one of three dose groups. Information about doses will be provided before the start of the vaccinations.
* Vaccine injections will be given at the start of the study, at 4 weeks, and at 20 weeks. Participants will be asked to keep an eye on the injection site for 7 days and to notify researchers if there are any side effects.
* Participants will be monitored throughout the study with blood samples and clinic visits.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation study to examine the safety, tolerability, and immune response to a Virus-Like Particle (VLP) Chikungunya Virus (CHIKV) vaccine in healthy adults ages 18 to 50 years old. The plan is for 25 subjects to receive 3 intramuscular vaccine injections at weeks 0, 4, and 20. The three groups will be enrolled sequentially starting with the lowest dose of 10 micrograms per injection in Group 1.

The hypothesis is that the vaccine is safe and induces immune responses to CHIKV. The primary objective is to evaluate the safety and tolerability of the investigational vaccine, VRC-CHKVLP059-00-VP, at three dosages, 10 micrograms (mcg), 20 mcg, and 40 mcg, in healthy adults. The secondary objective is to evaluate the antibody response against CHIKV VLPs four weeks after the third vaccine injection. The exploratory objectives relate to antigen-specific humoral and cellular immune responses throughout the study.

ELIGIBILITY:
INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 50 years old
2. Available for clinical follow-up through Week 44
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
4. Complete an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly
5. Able and willing to complete the informed consent process
6. Willing to donate blood for sample storage to be used for future research
7. In good general health, with a BMI less than or equal to 40, without clinically significant medical history, and has satisfactorily completed screening
8. Physical examination and laboratory results without clinically significant findings within the 56 days prior to enrollment

   Laboratory Criteria within 56 days prior to enrollment:
9. Hemoglobin greater than or equal to11.5 g/dL for women; greater than or equal to13.5 g/dL for men
10. WBC: 3,000-12,000 cells/mm(3).
11. Differential either within institutional normal range or accompanied by physician approval
12. Total lymphocyte count: greater than or equal to 800 cells/mm(3)
13. Platelets = 125,000-500,000/mm(3)
14. Alanine aminotransferase (ALT) less than or equal to 1.25 times upper limit of normal range
15. Serum creatinine less than or equal to1x upper limit of normal (less than or equal to1.3 mg/dL for females; less than or equal to1.4 mg/dL for males).
16. Negative FDA-approved HIV blood test

    Female-Specific Criteria
17. Negative Beta-HCG pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential
18. A woman of childbearing potential must agree to use an effective means of birth control from at least 21 days prior to enrollment through 12 weeks after last study vaccination

EXCLUSION CRITERIA:

A participant will be excluded if one or more of the following conditions apply:

Female-Specific Criteria

1. Woman who is breast-feeding or planning to become pregnant during the time projected for individual study participation
2. Systemic immunosuppressive medications or cytotoxic medications within 12 weeks prior to enrollment [with the exceptions that a short course of corticosteroids (less than or equal to10 days duration or a single injection) for a self-limited condition at least 2 weeks prior to enrollment will not exclude study participation]
3. Blood products within 16 weeks prior to enrollment
4. Immunoglobulin within 8 weeks prior to enrollment
5. Prior vaccinations with an investigational CHIKV vaccine
6. Investigational research agents within 4 weeks prior to enrollment
7. Live attenuated vaccines within 4 weeks prior to enrollment
8. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 2 weeks prior to enrollment
9. Current anti-TB prophylaxis or therapy

   Subject has a history of any of the following clinically significant conditions:
10. A history of confirmed or suspected CHIKV infection
11. A history of immune-mediated or clinically significant arthritis
12. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator
13. Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema
14. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that is expected to require the use of oral or intravenous corticosteroids
15. Diabetes mellitus (type I or II), with the exception of gestational diabetes
16. Idiopathic urticaria within the past year
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
18. Malignancy that is active, or treated malignancy for which there is not reasonable assurance of sustained cure, or malignancy that is likely to recur during the period of the study
19. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
20. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
21. Psychiatric condition that may preclude compliance with the protocol; past or present psychoses; disorder requiring lithium; or within five years prior to enrollment, a history of suicide plan or attempt
22. Any medical condition (such as thyroid disease or hypertension that are not well controlled by medication, or viral hepatitis) that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, D.O., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Strauss JH, Strauss EG. The alphaviruses: gene expression, replication, and evolution. Microbiol Rev. 1994 Sep;58(3):491-562. doi: 10.1128/mr.58.3.491-562.1994. PMID 7968923
- [Background] Powers AM, Logue CH. Changing patterns of chikungunya virus: re-emergence of a zoonotic arbovirus. J Gen Virol. 2007 Sep;88(Pt 9):2363-2377. doi: 10.1099/vir.0.82858-0. No abstract available. PMID 17698645
- [Background] Volk SM, Chen R, Tsetsarkin KA, Adams AP, Garcia TI, Sall AA, Nasar F, Schuh AJ, Holmes EC, Higgs S, Maharaj PD, Brault AC, Weaver SC. Genome-scale phylogenetic analyses of chikungunya virus reveal independent emergences of recent epidemics and various evolutionary rates. J Virol. 2010 Jul;84(13):6497-504. doi: 10.1128/JVI.01603-09. Epub 2010 Apr 21. PMID 20410280
- [Derived] Chang LJ, Dowd KA, Mendoza FH, Saunders JG, Sitar S, Plummer SH, Yamshchikov G, Sarwar UN, Hu Z, Enama ME, Bailer RT, Koup RA, Schwartz RM, Akahata W, Nabel GJ, Mascola JR, Pierson TC, Graham BS, Ledgerwood JE; VRC 311 Study Team. Safety and tolerability of chikungunya virus-like particle vaccine in healthy adults: a phase 1 dose-escalation trial. Lancet. 2014 Dec 6;384(9959):2046-52. doi: 10.1016/S0140-6736(14)61185-5. Epub 2014 Aug 14. PMID 25132507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited at the NIH Clinical Center in Bethesda, Maryland from December 12, 2011 to March 22, 2012
Groups:
- Group 1: 10 mcg VRC-CHKVLP059-00-VP: Group 1 subjects received 10 mcg of a Virus-Like Particle (VLP) Chikungunya Vaccine, VRC-CHKVLP059-00-VP, on Days 0, 28, and 140
- Group 2: 20 mcg VRC-CHKVLP059-00-VP: Group 2 subjects received 20 mcg of a Virus-Like Particle (VLP) Chikungunya Vaccine, VRC-CHKVLP059-00-VP, on Days 0, 28, and 140
- Group 3: 40 mcg VRC-CHKVLP059-00-VP: Group 3 subjects received 40 mcg of a Virus-Like Particle (VLP) Chikungunya Vaccine, VRC-CHKVLP059-00-VP, on Days 0, 28, and 140
Period: Overall Study
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Started | 5 | 10 | 10
Completed | 5 | 10 | 8
Not Completed | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP | Total
Number analyzed (Participants) | 5 | 10 | 10 | 25
Age, Customized [Number; unit: participants]
  18-20 years | 1 | 0 | 0 | 1
  21-30 years | 2 | 4 | 6 | 12
  31-40 years | 2 | 4 | 3 | 9
  41-50 years | 0 | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 10
  Male | 2 | 7 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 3 | 8 | 8 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of First Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after first vaccination and review the Memory Aid with clinic staff at follow a up visit. Subjects are counted once for each symptom if they indicated experiencing the symptom at any severity during the reporting period. The number reported for all local symptoms is the number reporting one or more local symptom at any severity.
Time Frame: 7 days after the first vaccination
Population: All subjects who received the first vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants
  Pain/Tenderness | 0 | 1 | 1
  Swelling | 0 | 0 | 0
  Redness | 0 | 0 | 0
  Any Local Symptom | 0 | 1 | 1

2. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Second Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after second vaccination and review the Memory Aid with clinic staff at follow a up visit. Subjects are counted once for each symptom if they indicated experiencing the symptom at any severity during the reporting period. The number reported for all local symptoms is the number reporting one or more local symptom at any severity.
Time Frame: 7 days after the second vaccination
Population: All subjects who received the second vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants
  Pain/Tenderness | 0 | 2 | 3
  Swelling | 0 | 0 | 0
  Redness | 0 | 0 | 0
  Any Local Symptom | 0 | 2 | 3

3. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Third Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after third vaccination and review the Memory Aid with clinic staff at follow a up visit. Subjects are counted once for each symptom if they indicated experiencing the symptom at any severity during the reporting period. The number reported for all local symptoms is the number reporting one or more local symptom at any severity.
Time Frame: 7 days after the third vaccination
Population: Number of subjects who received the third vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 8
participants
  Pain/Tenderness | 1 | 3 | 4
  Swelling | 0 | 0 | 0
  Redness | 0 | 0 | 0
  Any Local Symptom | 1 | 3 | 4

4. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Any Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after any vaccination and review the Memory Aid with clinic staff at follow a up visit. Subjects are counted once for each symptom if they indicated experiencing the symptom at any severity during the reporting period. The number reported for all local symptoms is the number reporting one or more local symptom at any severity.
Time Frame: 7 days after any vaccination
Population: Number of subjects who received at least one vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants
  Pain/Tenderness | 1 | 4 | 4
  Swelling | 0 | 0 | 0
  Redness | 0 | 0 | 0
  Any Local Symptom | 1 | 4 | 4

5. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of First Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after first vaccination and review the Memory Aid with clinic staff at follow a up visit. Subjects are counted once for each symptom if they indicated experiencing the symptom at any severity during the reporting period. The number reported for all systemic symptoms is the number reporting one or more systemic symptom at any severity.
Time Frame: 7 days after the first vaccination
Population: All subjects who received the first vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants
  Malaise | 1 | 1 | 1
  Myalgia | 0 | 0 | 1
  Headache | 0 | 0 | 1
  Chills | 0 | 0 | 0
  Nausea | 0 | 0 | 2
  Temperature | 0 | 0 | 0
  Joint Pain | 0 | 0 | 0
  Any Systemic Symptom | 1 | 1 | 3

6. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Second Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after second vaccination and review the Memory Aid with clinic staff at follow a up visit. Subjects are counted once for each symptom if they indicated experiencing the symptom at any severity during the reporting period. The number reported for all systemic symptoms is the number reporting one or more systemic symptom at any severity.
Time Frame: 7 days after the second vaccination
Population: All subjects who received the second vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants
  Malaise | 0 | 1 | 0
  Myalgia | 0 | 1 | 0
  Headache | 0 | 0 | 1
  Chills | 0 | 0 | 0
  Nausea | 1 | 0 | 1
  Temperature | 0 | 0 | 0
  Joint Pain | 0 | 0 | 0
  Any Systemic Symptom | 1 | 1 | 2

7. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Third Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after third vaccination and review the Memory Aid with clinic staff at follow a up visit. Subjects are counted once for each symptom if they indicated experiencing the symptom at any severity during the reporting period. The number reported for all systemic symptoms is the number reporting one or more systemic symptom at any severity.
Time Frame: 7 days after the third vaccination
Population: Number of subjects who received the third vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 8
participants
  Malaise | 0 | 2 | 1
  Myalgia | 0 | 1 | 0
  Headache | 1 | 0 | 1
  Chills | 0 | 0 | 0
  Nausea | 0 | 0 | 1
  Temperature | 0 | 0 | 0
  Joint Pain | 0 | 0 | 0
  Any Systemic Symptom | 1 | 2 | 2

8. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Any Vaccination
Description: Subjects record the occurrence of solicited symptoms on a Memory Aid for 7 days after any vaccination and review the Memory Aid with clinic staff at follow a up visit. Subjects are counted once for each symptom if they indicated experiencing the symptom at any severity during the reporting period. The number reported for all systemic symptoms is the number reporting one or more systemic symptom at any severity.
Time Frame: 7 days after any vaccination
Population: All subjects who received at least one vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants
  Malaise | 1 | 3 | 2
  Myalgia | 0 | 2 | 1
  Headache | 1 | 0 | 3
  Chills | 0 | 0 | 0
  Nausea | 1 | 0 | 3
  Temperature | 0 | 0 | 0
  Joint Pain | 0 | 0 | 0
  Any Systemic Symptom | 2 | 3 | 5

9. Primary Outcome: Number of Subjects With an Any Abnormal Laboratory Result
Description: Blood samples were collected for chemistry, CBC with differential, at baseline and weeks 2, 4, 6, 8, 20, 22, 24 and 44
Time Frame: 44 weeks after first vaccination
Population: All subjects who received at least one vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants
  ALT | 1 | 2 | 2
  WBC | 3 | 3 | 0
  Hemoglobin | 1 | 2 | 1
  Platelets | 0 | 0 | 0
  Neutrophil Count | 2 | 1 | 2
  Lymphocyte Count | 1 | 1 | 0
  Eosinophil Count | 1 | 1 | 1
  Any Abnormal Lab Result | 4 | 5 | 5

10. Primary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events were collected at each study visit from the time of first vaccination through the final study visit at 44 weeks after the first vaccination.
Time Frame: 44 weeks after first vaccination
Population: All subjects who received at least one vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants | 0 | 0 | 0

11. Primary Outcome: Number of Subjects Reporting 1 or More Unsolicited Adverse Event
Description: Unsolicited adverse events were recorded from enrollment through 28 days after the second vaccination; and from the third vaccination through 28 days after this vaccination.
  Between and after the indicated time periods, through the last expected study visit (i.e., 24 weeks after the third vaccination), only SAEs and new chronic medical conditions were recorded. The number of unsolicited events reported for Group 3 here is lower than the total number of adverse events in the Adverse Event Module, which reports both solicited and unsolicited adverse events.
Time Frame: 28 days after each vaccination
Population: All subjects who received at least one vaccination
Measure: Number; unit: participants
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
participants
  Any AE | 4 | 9 | 6
  Blood and Lymphatic System Disorders | 2 | 2 | 1
  Infections and Infestations | 3 | 5 | 4
  Injury, Poisoning and Procedural Complications | 0 | 2 | 0
  Investigations | 1 | 0 | 2
  Musculoskeletal and Connective Tissue Disorders | 1 | 1 | 0
  Surgical and Medical Procedures | 0 | 0 | 1
  Vascular Disorders | 0 | 1 | 0

12. Secondary Outcome: Chikungunya Antigen-specific ELISA Geometric Mean Titer (GMT)
Description: ELISA titer (strain 37997) For ELISA, week 0 values were used to background correct titres for subsequent weeks.
Time Frame: 24 weeks after the first vaccination
Population: All subjects who received at least one vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titre
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
titre | 40960 [40960 to 40960] | 15521 [6058 to 39763] | 34443 [22862 to 51890]

13. Secondary Outcome: Chikungunya Antigen-specific Neutralizing Antibody Geometric Mean Titer (GMT)
Description: Neutralisation IC50 titre (strain OPY1)
Time Frame: Pre-vaccination (Week 0)
Population: All subjects who received at least one vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titre
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
titre | 50 [50 to 50] | 51 [49 to 52] | 52 [50 to 54]

14. Secondary Outcome: Chikungunya Antigen-specific Neutralizing Antibody Geometric Mean Titer (GMT)
Description: Neutralisation IC50 titre (strain OPY1)
Time Frame: 24 weeks after the first vaccination
Population: All subjects who received at least one vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titre
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Number analyzed (Participants) | 5 | 10 | 10
titre | 8745 [1514 to 50516] | 4525 [2252 to 9093] | 5390 [1865 to 15573]

ADVERSE EVENTS:
Time Frame: Solicited symptoms collected 7 days after each vaccination; unsolicited non-serious, non-chronic adverse events, through 28 days after each vaccination; Serious adverse events and new chronic medical conditions, through 24 weeks after last vaccination.
Description: For the solicited symptoms, participants are counted if reporting the symptom after any vaccination, with the occurrence within 0-7 days of a vaccination considered 1 event.
Arm/Group | Group 1: 10 mcg VRC-CHKVLP059-00-VP | Group 2: 20 mcg VRC-CHKVLP059-00-VP | Group 3: 40 mcg VRC-CHKVLP059-00-VP
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/5 | 9/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 10 mcg VRC-CHKVLP059-00-VP (N=5) | Group 2: 20 mcg VRC-CHKVLP059-00-VP (N=10) | Group 3: 40 mcg VRC-CHKVLP059-00-VP (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 2
Viral Infection (Infections and infestations) | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Incisional drainage (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Pain/Tenderness (General disorders) | 1 | 4 | 4
Headache (Nervous system disorders) | 1 | 0 | 3
Malaise (General disorders) | 1 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes